CLINICAL TRIAL: NCT02328209
Title: Evaluation of the Efficacy and Continuance Rate of Treatment in Simplified Treat And Extend Regimen Using Ranibizumab in Exudative Age Related Macular Degeneration
Brief Title: Evaluation of the Simplified Treat And Extend Regimen Using Ranibizumab in Exudative Age Related Macular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mie University (Other)
Responsible Party: Principal Investigator, Mineo Kondo, Mie University Graduate School of Medicine, Mie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000014056
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Exudative Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ranibizumab (Experimental): ranibizumab
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg/0.05ml, intravitreal injection, frequency: each 8 or 12 weeks
  Other Names: Lucentis

SUMMARY:
Recently studies have shown that intravitreal injection of ranibizumab is effective for age related macular degeneration. However there are problems about injection regimen of maintenance phase. We plan to perform new simplified treat and extend regimen using ranibizumab.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate the simplified treat and extend regimen using ranibizumab in eyes with wet age related macular degeneration about best-corrected visual acuity, central retinal thickness, the disappearance rate of the morphological change and treatment continuous rate.

ELIGIBILITY:
Inclusion Criteria:

1. ability to provide written informed consent for this study
2. age>=50years old
3. intravitreal injection of ranibizumab as a first therapy for neovascular age-related macular degeneration (typical age-related macular degeneration and PCV)
4. best corrected visual acuity>=0.05 -

Exclusion Criteria:

1. past intravitreal anti-vascular endothelial growth factor therapy in the study eye
2. past intravitreal or subtenon injection of steroid therapy in the study eye
3. past vitrectomy therapy in the study eye
4. infection or suspicion of infection in eyes or periocular region
5. severe intraocular inflammation in eyes
6. past allergic reaction for ranibizumab
7. past allergic reaction for fluorescein, indocyanine green or iodine
8. pregnancy (positive pregnancy test) or lactating women
9. other conditions that the investigator believed would pose a significant hazard to the subject if investigational therapy were initiated.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
A change from baselines best corrected visual acuity at 24 months | 24 months

SECONDARY OUTCOMES:
A drop-out rate of the 3 and 12 months | 3 and 12 months
A treatment continuance rate until 24 months | 24 months
A change of best corrected visual acuity at 12 months | 12 months
A change from baselines central retinal thickness measured by spectral domain optical coherence tomography at 12 and 24 months | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mineo Kondo, Study Chair — Mie University
Locations (1):
- Mie University Graduate School of Medicine, Tsu, Japan

REFERENCES:
- [Result] Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP, Schneider S; ANCHOR Study Group. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1432-44. doi: 10.1056/NEJMoa062655. PMID 17021319
- [Result] Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY, Kim RY; MARINA Study Group. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006 Oct 5;355(14):1419-31. doi: 10.1056/NEJMoa054481. PMID 17021318